CLINICAL TRIAL: NCT06344325
Title: 90% Effective Dose Study of Fospropofol Disodium in Induction and Maintenance of Anesthesia in Adults of Different Ages
Brief Title: ED90 of Fospropofol Disodium in Induction and Maintenance of Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Clinical Professor, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EDPP
Record Dates: First submitted 2024-03-26; First posted 2024-04-03 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Elective Surgery
MeSH Terms: interventions — fospropofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Youth group (Experimental): Youth group (18-45 years old)
  Interventions: Drug: fospropofol
- middle-aged group (Experimental): middle-aged group (46-65 years old)
  Interventions: Drug: fospropofol
- elderly group (Experimental): elderly group (66-80 years old)
  Interventions: Drug: fospropofol

INTERVENTIONS:
Drug: fospropofol — The initial dose of fospropofol disodium in the youth group is 15mg/kg,the middle-aged group is 10mg/kg, the elderly group is 7.5mg/kg, and the concentration of adjacent intervals is 0.5mg/kg.
  Other Names: fospropofol disodium

SUMMARY:
Exploring the 90% effective dose (ED90) of fospropofol disodium in induction and maintenance of anesthesia in adults of different ages, providing more clinical evidence for the application of fospropofol disodium in clinical anesthesia

DETAILED DESCRIPTION:
As a newly marketed sedative hypnotic agent, fospropofol disodium is currently the only water-soluble precursor drug of propofol in China. It has the characteristics of long duration of action, low incidence of injection pain, respiratory and circulatory system related adverse events, and no lipid metabolism related adverse reactions, providing anesthesiologists with another sedative option during surgery. However, there are currently few clinical observation studies on this drug, and there have been no reports on its effective dosage in different age groups. Therefore, this study aims to observe the 90% effective dose (ED90) in anesthesia induction and maintenance in adults of different ages, providing effective clinical evidence for its application in clinical anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years old, elective surgery under general anesthesia.
* ASA I-II;
* Surgical duration>30 minutes;
* Sign an informed consent form.

Exclusion Criteria:

* American Society of Anesthesiologists(ASA)≥ III;
* Body mass index (BMI)<18 kg/m2 or>30 kg/m2;
* Individuals with a history or potential history of drug abuse or alcohol dependence;
* Preoperative use of sedative or analgesic drugs;
* Individuals with severe liver and kidney dysfunction;
* Individuals who are allergic or potentially allergic to propofol and lipids;
* The types of surgeries that directly affect hemodynamics, such as large vessel surgery and other surgical procedures;
* Patients with abnormal coagulation function, endocrine disorders, or other factors affecting hemodynamic status;
* Participants in other clinical studies within the past 3 months;
* researchers deemed it inappropriate for participants to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Sedation score | 1 day
  Sedation score (MOAA/S)

SECONDARY OUTCOMES:
Postoperative adverse reactions | 1 day
  Postoperative adverse reactions such as Hypertension, hypotension, tachycardia, gastrointestinal symptoms, postoperative restlessness.

CONTACTS AND LOCATIONS:
Overall Officials: aihua Du, Dr., Study Chair — Tongji Hospital
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No